CLINICAL TRIAL: NCT04266262
Title: High-Intensity Training for Men With Prostate Cancer on Active Surveillance: A Feasibility Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: All research activities were suspended as a result of COVID-19.
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Daniel Santa Mina, PhD, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-6340
Record Dates: First submitted 2020-02-06; First posted 2020-02-12 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
Keywords: Active Surveillance; Prostate Cancer; High-intensity interval training; Resistance training
MeSH Terms: conditions — Prostatic Neoplasms | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Intensity interval training (HIIT) (Experimental)
  Interventions: Behavioral: High-intensity interval training (HIIT)
- High-intensity resistance training (HIRT) (Experimental)
  Interventions: Behavioral: High-Intensity resistance training (HIRT)
- Usual care (UC) (No Intervention): Provision of Cancer Care Ontario's physical activity guidelines for cancer survivors

INTERVENTIONS:
Behavioral: High-intensity interval training (HIIT) — Supervised HIIT sessions (2x/week) will comprise cycling 10 x 60 secs at 85-95% maximum heart rate (HRmax) interspersed by 60 secs of low-intensity recovery.
  Unsupervised HIIT sessions (1x/week) will involve 10 x 60 secs of walking or alternative (intensity of 7-9 on the 0-10 RPE) interspersed by 60 secs of walking or cycling at low intensity recovery (RPE 3-5).
  Arms: High-Intensity interval training (HIIT)
Behavioral: High-Intensity resistance training (HIRT) — Supervised HIRT sessions (2x/week) will comprise 2-3 sets of 6-8 repetitions progressively achieving 85% of 1RM.
  Unsupervised HIRT sessions (1x/week) will involve 2-3 sets of 15-20 repetitions using a resistance exercise band when necessary.
  Arms: High-intensity resistance training (HIRT)

SUMMARY:
This is a randomized study aiming to assess the feasibility of a phase II randomized controlled trial of different high-intensity training interventions and usual care (UC) in men with prostate cancer (PCa) undergoing active surveillance (AS).

DETAILED DESCRIPTION:
Primary objectives:

The primary objective of this study is to assess the feasibility of conducting a three-armed randomized controlled trial comparing high-intensity interval training (HIIT), high-intensity resistance training (HIRT), and usual care (UC) in men with PCa on AS.

The secondary exploratory objective of this study is to assess changes in cardiorespiratory fitness, musculoskeletal strength, body composition, circulating blood markers, and participant-self-reported outcomes (e.g., quality of life, anxiety, fear of disease progression) after 8 weeks of HIIT, HIRT, or UC.

Methods:

Participants will be randomized in a 1:1:1 ratio to HIIT, HIRT or UC group.

Participants in the HIIT and HIRT group will undergo training 3 times per week (two supervised and one home-based/unsupervised training session) for 8 weeks.

The UC group will be directed towards publicly available literature on physical activity (e.g., Cancer Care Ontario's physical activity guidelines for cancer survivors) and will receive an individualized exercise program upon completion of their final fitness assessment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* initiating or currently on AS for PCa;
* not currently engaging in high-intensity aerobic and/or resistance training at 85%HRmax or ≥9 RPE in the Borg 0-10 RPE scale;
* willing and able to travel to the study-designated facilities;
* proficient in English;
* able to provide written informed consent;
* pass the screening CPET by achieving volitional exhaustion (rate of perceived exertion (RPE) ≥ 9 using the Borg 0-10 RPE scale) in the absence of any cardiorespiratory abnormalities.

Exclusion Criteria:

* uncontrolled hypertension (≥2/3 of readings of > 160/90), regardless of whether on a regimen of anti-hypertensive therapy or not;
* been diagnosed with congestive heart failure (New York Heart Association Class II, III or IV);
* a history of serious cardiovascular events (within 12 months) including, but not limited to, transient ischemic attack (TIA), cerebrovascular accident (CVA), or myocardial infarction (MI);
* a medical condition such as uncontrolled infection or cardiac disease that, in the opinion of the study physician, would make this protocol unreasonably hazardous for the patient;
* a history of a psychiatric illness, which would prevent the patient from giving informed consent or adhering to the study protocol;
* serious or non-healing wound, ulcer, or bone fracture;
* experience shortness of breath, chest discomfort, or palpitations when performing activities of daily living;
* ongoing restriction of physical activity;
* developed chest pain in the past month

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Recruitment rate (feasibility target: ≥25% of eligible patients) | Initiation through end of study recruitment at 26 months
  Percent of consenting participants relative to the total number of eligible participants approached
Attendance rate (feasibility target: ≥70% to facility-based sessions) | Initiation through end of study intervention period at a maximum of 8 weeks post-randomization
  Percent of completed facility-based sessions relative to the total number of prescribed facility-based sessions
Compliance rate (feasibility target: ≥70% of the prescribed exercises within supervised sessions) | Initiation through end of study intervention period at a maximum of 8 weeks post-randomization
  Percent of completed repetitions relative to the total number of prescribed repetitions
Retention rate (feasibility target: 70% of participants consented to study) | Initiation through end of study intervention period at a maximum of 8 weeks post-randomization
  Percent of participants that completed the study relative to the total number of participants consented to the study

SECONDARY OUTCOMES:
Changes in cardiorespiratory fitness | At baseline and 8 weeks (post-intervention)
  Cardiopulmonary exercise test (CPET)-based assessment of peak oxygen uptake (VO2peak)
Changes in musculoskeletal strength | At baseline and 8 weeks (post-intervention)
  1 repetition maximum (1RM) will be assessed for upper (e.g., seated row and chest press) and lower body (e.g., leg press)
Changes in circulating cytokines | At baseline and 8 weeks (post-intervention)
  TNFalpha, interleukin (IL)-6, and IL-10 will be assessed using blood samples
Changes in circulating growth factors | At baseline and 8 weeks (post-intervention)
  Insulin-like growth factor-1 (IGF-1) and insulin-like binding protein 3 (IGFBP-3) will be assessed using blood samples
Body composition | At baseline and 8 weeks (post-intervention)
  Body mass will be measured using a weight scale (kg)
Changes in waist circumference | At baseline and 8 weeks (post-intervention)
  Waist circumference will be measured using a measuring tape (cm)
Changes in body fat and lean body mass | At baseline and 8 weeks (post-intervention)
  % body fat and % lean body mass will be measured using a bioelectrical impedance analysis (BIA) scale
Changes in Quality of Life | At baseline and 8 weeks (post-intervention)
  QoL will be measured using the Functional Assessment of Cancer Therapy-Prostate (FACT-P)
Anxiety | At baseline and 8 weeks (post-intervention)
  Anxiety will be measured using the Hospital Anxiety and Depression Scale (HADS) and the Memorial Anxiety Scale for Prostate Cancer (MAX-PC)
Fear of disease progression | At baseline and 8 weeks (post-intervention)
  Fear of disease progression will be measured using the Fear of Progression Questionnaire-Short Form (FOP-Q-SF)
Physical activity status | At baseline and 8 weeks (post-intervention)
  Changes in physical activity status will be measured using the Godin-Leisure Time Physical Activity Questionnaire (GLTEQ)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data of this study will be available from the corresponding author upon reasonable request

REFERENCES:
- [Derived] Papadopoulos E, Gillen J, Moore D, Au D, Kurgan N, Klentrou P, Finelli A, Alibhai SMH, Santa Mina D. High-intensity interval training or resistance training versus usual care in men with prostate cancer on active surveillance: a 3-arm feasibility randomized controlled trial. Appl Physiol Nutr Metab. 2021 Dec;46(12):1535-1544. doi: 10.1139/apnm-2021-0365. Epub 2021 Aug 11. PMID 34380000